CLINICAL TRIAL: NCT02604901
Title: Effect of Community Pharmacist Intervention on Adherence to Long-Term Medications
Acronym: ECO-PHIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Rite Aid Corp. (Industry); RTI International (Other); Pharmacy Quality Alliance (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jan Pringle, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: ECOPHIL
Record Dates: First submitted 2015-11-05; First posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Medication Adherence
Keywords: medication adherence; community pharmacies; screening and brief intervention
MeSH Terms: conditions — Medication Adherence | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Screening and Brief Intervention (BI) (Experimental): Screening and Brief Intervention (BI) at initial prescription fill and at each additional refill.
  Interventions: Behavioral: Screening and Brief Intervention (BI)
- Pill Box (PB) (Experimental): Pill Box (PB) and information about their medications at the initial fill and at each additional refill.
  Interventions: Behavioral: Pill Box (PB)
- Brief Intervention + Pill Box (BI+PB) (Experimental): Screening and Brief Intervention (BI) and Pill Box (PB) at initial prescription fill and at each additional refill.
  Interventions: Behavioral: Screening and Brief Intervention (BI); Behavioral: Pill Box (PB)
- Standard Care (SC) (No Intervention): The Standard Care (SC) arm administered traditional dispensing and counseling by Rite Aid® pharmacists.

INTERVENTIONS:
Behavioral: Screening and Brief Intervention (BI) — Rite Aid® pharmacists screened patients at the time of the initial fill with the Adherence Estimator™ and using the screening results, provided the behavioral intervention, Brief Intervention using motivational interviewing principles based on POLAR*S (BI). BI was considered an active intervention method.
  Arms: Brief Intervention + Pill Box (BI+PB); Screening and Brief Intervention (BI)
Behavioral: Pill Box (PB) — Rite Aid® pharmacists provided patients with a Pill Box (PB) and information about their medications. However, pharmacists did not use motivational interviewing principles for engaging patients in direct interventions to modify behavior. PB was considered a passive intervention method.
  Arms: Brief Intervention + Pill Box (BI+PB); Pill Box (PB)

SUMMARY:
The 4-arm factorial design RCT tested the impact of a behavioral intervention (SBI or BI), a reminder device (Pillbox), and the combination of the two on adherence in adult patients who filled a prescription for oral medications to treat diabetes or hyperlipidemia.

DETAILED DESCRIPTION:
Patients diagnosed with chronic diseases often fail to follow their prescribed medication regimens, (16355071,19954264,16732693,23111664) which accounts for up to 290 billion dollars per year in unnecessary medical costs, largely because medication nonadherence increases their risk of disease progression, hospitalization, and premature death.(16355071, 23373139, 23032359) A number of studies have investigated ways to improve medication adherence; (18425859, 18537843) however, few studies on interventions have demonstrated large improvements in adherence and few have used scientifically rigorous study methods such as randomized controlled trials (RCTs).(24422970) A recent systematic review identified a need for adherence interventions and suggested the use of factorial designs in RCTs to study multiple interventions and combinations within large patient populations.(24422970)

This study used a factorial-designed, four-armed, RCT to examine the impact of three pharmacy-based interventions versus standard care on improving medication adherence and health outcomes in patients with diabetes and hyperlipidemia. The three interventions used in this study were a behavioral intervention, a pillbox weekly reminder, and the combination of the two.

Pillboxes (PB) used in this study had compartments for each day (7X1) and for participants taking multiple medications, sub-compartments for each medication per day (7X4).

The behavioral intervention, called Screening and Brief Intervention (SBI or BI), consisted of a short 2-5 minute conversation between the patient and the provider aimed to encourage modification in the patient's health behavior. While BI has primarily been used to address unhealthy alcohol use in patients (11), the researchers hypothesized that this patient-centered approach can be particularly useful for improving medication adherence in chronically ill patients. In this study, motivational interviewing counseling principles were used for motivating patients to take more active roles in self-managing their health. Motivational interviewing can take many forms, however, in this study, the BIs used a schema of motivational interviewing originally developed by the principal investigator titled POLAR*S™ .

The specific aims of this research study included testing the impact of three community pharmacy intervention for adult patients with diabetes or hyperlipidemia on: (1) medication adherence; (2) biologic outcomes associated with medication adherence; (3) self-reported health and psychosocial status; and (4) pharmacists' impressions on how BI could be scalable to community pharmacy settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients taking oral medications for diabetes or hyperlipidemia
* 30-85 years of age
* Comfortable speaking in English
* Not institutionalized
* Not diagnosed with psychosis or dementia.
* Needed at least one prescription refill with the index medication picked up within 14 days of the index prescription fill

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1091 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence using the PDC metric, for adult patients with diabetes or hyperlipidemia. | At baseline and nine-months post-enrollment into the study.
  Medication adherence was measured as a Proportion of Days Covered (PDC) by calculating (at the patient level) the denominator as the number of days between the first fill of the medication during a measurement period and the end of the measurement period and the numerator is calculated as the number of days covered by prescription fill date and days of supply. For each patient, the PDC was calculated at baseline and 9-months. The baseline PDC was compared to that at 9-months.

SECONDARY OUTCOMES:
Change in triglyerceride levels from baseline to 6- and 9-months. | At baseline, six months and nine-months post-enrollment into the study.
  Triglyeride levels were measured for patients who had regular blood samples drawn, at baseline, 6-months, and 9-months, by their physician during the course of the study. The baseline measure was compared to that at 6- and 9-months.
Change in cholesterol levels from baseline to 6- and 9-months. | At baseline, six months and nine-months post-enrollment into the study.
  Cholesterol levels were measured for patients who had regular blood samples drawn, at baseline, 6-months, and 9-months, by their physician during the course of the study. The baseline measure was compared to that at 6- and 9-months.
Change in high-density lipoprotein (HDL) levels from baseline to 6- and 9-months. | At baseline, six months and nine-months post-enrollment into the study.
  High-density lipoprotein (HDL) levels were measured for patients who had regular blood samples drawn, at baseline, 6-months, and 9-months, by their physician during the course of the study. The baseline measure was compared to that at 6- and 9-months.
Change in low-density lipoprotein (LDL) levels from baseline to 6- and 9-months. | At baseline, six months and nine-months post-enrollment into the study.
  Low-density lipoprotein (LDL) levels were measured for patients who had regular blood samples drawn, at baseline, 6-months, and 9-months, by their physician during the course of the study. The baseline measure was compared to that at 6- and 9-months.
Change in glycated hemoglobin (HbA1c) levels from baseline to 6- and 9-months. | At baseline, six months and nine-months post-enrollment into the study.
  Glycated hemoglobin (HbA1c) levels were measured for patients who had regular blood samples drawn, at baseline, 6-months, and 9-months, by their physician during the course of the study. The baseline measure was compared to that at 6- and 9-months.
Change in self-reported healthcare utilization, using a study-designed standardized questionnaire, from baseline to 9-months. | At baseline and nine-months post-enrollment into the study.
  Self-reported healthcare utilization information was collected upon enrollment during the baseline interview using a standardized questionnaire developed bv the PI for the study. These interviews were repeated for the 9-month follow-up period.
Change in self-reported psychosocial status, using a study-designed standardized questionnaire, from baseline to 9-months. | At baseline and nine-months post-enrollment into the study.
  Self-reported psychosocial status information was collected upon enrollment during the baseline interview using a standardized questionnaire developed bv the PI for the study. These interviews were repeated for the 9-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Janice L Pringle, PhD, Principal Investigator — University of Pittsburgh; Newell McElwee, PharmD, MSPH, Study Chair — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Rite Aid® Corporation, Marietta, Georgia
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Yeaw J, Benner JS, Walt JG, Sian S, Smith DB. Comparing adherence and persistence across 6 chronic medication classes. J Manag Care Pharm. 2009 Nov-Dec;15(9):728-40. doi: 10.18553/jmcp.2009.15.9.728. PMID 19954264
- [Background] Vik SA, Hogan DB, Patten SB, Johnson JA, Romonko-Slack L, Maxwell CJ. Medication nonadherence and subsequent risk of hospitalisation and mortality among older adults. Drugs Aging. 2006;23(4):345-56. doi: 10.2165/00002512-200623040-00007. PMID 16732693
- [Background] Traynor K. Poor medication adherence remains a problem. Am J Health Syst Pharm. 2012 Nov 1;69(21):1850. doi: 10.2146/news120074. No abstract available. PMID 23111664
- [Background] Stefanacci RG, Guerin S. Why medication adherence matters to patients, payers, providers. Manag Care. 2013 Jan;22(1):37-9. No abstract available. PMID 23373139
- [Background] Williams J, Steers WN, Ettner SL, Mangione CM, Duru OK. Cost-related nonadherence by medication type among Medicare Part D beneficiaries with diabetes. Med Care. 2013 Feb;51(2):193-8. doi: 10.1097/MLR.0b013e318270dc52. PMID 23032359
- [Background] Haynes RB, Ackloo E, Sahota N, McDonald HP, Yao X. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD000011. doi: 10.1002/14651858.CD000011.pub3. PMID 18425859
- [Background] Williams A, Manias E, Walker R. Interventions to improve medication adherence in people with multiple chronic conditions: a systematic review. J Adv Nurs. 2008 Jul;63(2):132-43. doi: 10.1111/j.1365-2648.2008.04656.x. PMID 18537843
- [Background] Viswanathan M, Golin CE, Jones CD, Ashok M, Blalock S, Wines RC, Coker-Schwimmer EJ, Grodensky CA, Rosen DL, Yuen A, Sista P, Lohr KN. Closing the quality gap: revisiting the state of the science (vol. 4: medication adherence interventions: comparative effectiveness). Evid Rep Technol Assess (Full Rep). 2012 Sep;(208.4):1-685. PMID 24422970
- [Background] Babor TF, Kadden RM. Screening and interventions for alcohol and drug problems in medical settings: what works? J Trauma. 2005 Sep;59(3 Suppl):S80-7; discussion S94-100. doi: 10.1097/01.ta.0000174664.88603.21. PMID 16355071